CLINICAL TRIAL: NCT07037069
Title: Effectiveness of Desensitization Training vs Graded Motor Imagery Training on Wrist Pain and Function in Patients With Reflex Sympathetic Dystrophy
Brief Title: Effectiveness of DT vs GMIT on Wrist Pain and Function in Patients With Reflex Sympathetic Dystrophy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1004
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Sympathetic; Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desensitization Training Group (Experimental)
  Interventions: Combination Product: Desensitization Training
- Graded Motor Imagery (GMI) (Experimental)
  Interventions: Combination Product: Graded Motor Imagery (GMI)

INTERVENTIONS:
Combination Product: Desensitization Training — Participants in this group received desensitization training aimed at reducing hypersensitivity and pain perception through progressive exposure to different tactile stimuli. Use of soft and coarse textures (cotton, wool, Velcro, brush). Rubbing, tapping, rolling over the affected wrist and hand.
  Arms: Desensitization Training Group
Combination Product: Graded Motor Imagery (GMI) — Training Sample Size: 20 participants Participants underwent a progressive 3-phase motor training program designed to target cortical reorganization and improve movement without provoking pain. Phases: Laterality Recognition - identifying left/right hand images (Recognise™ app or cards). Explicit Motor Imagery - visualizing wrist movements without actual motion. Mirror Therapy - using a mirror box to simulate movement of the affected wrist. Sessions: 30-45 minutes/day, 5 times/week, for 4 weeks.
  Arms: Graded Motor Imagery (GMI)

SUMMARY:
This study evaluated the effectiveness of two therapeutic approaches-Desensitization Training (DT) and Graded Motor Imagery (GMI)-in reducing wrist pain and improving function in patients with Reflex Sympathetic Dystrophy (RSD). The sample size was calculated using Epitools for one-way ANOVA comparison with two independent groups. A total of 40 participants were randomly assigned into two groups: the DT group and the GMI group, each consisting of 20 patients. The DT group underwent sessions involving progressive tactile stimulation using different textures and temperatures to reduce hypersensitivity and allodynia.

DETAILED DESCRIPTION:
In contrast, the GMI group followed a structured three-phase cognitive rehabilitation protocol including laterality recognition, explicit motor imagery, and mirror therapy, aimed at re-training cortical representation and reducing pain perception. Both groups received same number of sessions. Visual Analogue Scale (VAS), Patient Rated Wrist Evaluation (PRWE) & Specific Questionnaire for two groups is used to for pain and functional assessment involving wrist

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 65 years.
* Participants must have a confirmed diagnosis of Reflex Sympathetic Dystrophy (CRPS) Type I, affecting the wrist, according to the Budapest Criteria.
* Participants must experience chronic wrist pain for at least 3 months but not more than 24 months.
* Participants must be able to offer written informed consent and participate in the study willingly.
* Participants must demonstrate sufficient cognitive function to understand the training protocols (assessed via screening tools such as the Mini-Mental State Examination).

Exclusion Criteria:

* Participants who have undergone any surgical intervention for the wrist (other than the injury that led to RSD), or those with traumatic injuries that cause structural damage will be excluded.
* Participants with significant neurological disorders affecting the upper limb.
* Individuals with active psychiatric conditions, such as severe depression, anxiety, or psychosis which may impair participation in the study.
* Participants with poorly controlled medical conditions such as diabetes, cardiovascular disease, or autoimmune disorders that could interfere with treatment outcomes or the ability to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 6 Month
  A Visual Analogue Scale (VAS) is a measurement tool used to assess subjective characteristics, like pain intensity. It typically involves a 10 cm line with endpoints labeled "no pain" and "worst pain imaginable". The patient marks a point on the line that represents their pain level, and the score is determined by measuring the distance in millimeters (0-100) from the "no pain" end. VAS scores are commonly categorized as: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Patient-Rated Wrist Evaluation (PRWE) | 6 Months
  The Patient-Rated Wrist Evaluation (PRWE) is a 15-item questionnaire designed to assess pain and functional disability in individuals with wrist problems. It consists of two modules: a pain module with 5 items and a function module with 10 items, each scored on a scale of 0 to 10. The PRWE provides a way for patients to self-report their experiences with wrist pain and its impact on their daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- Hameed Latif Hospital Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No